CLINICAL TRIAL: NCT07313410
Title: Near-Infrared Diffuse Correlation Spectroscopy to Better Define the Pathophysiology of Peripheral Artery Disease
Brief Title: Using Near-Infrared Light to Better Understand Peripheral Artery Disease
Status: Recruiting | Type: Observational
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Michael Nelson, Professor, The University of Texas at Arlington
Other Study IDs: 2025-0414; 25CSA1432263 (Other Grant/Funding Number: AHA)
Record Dates: First submitted 2025-08-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Exercise MRI; Functional Performance; Ankle-Brachial Index; Questionnaires; MRI; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Plasma and Serum will be retained for up to 2 years after study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Individuals without PAD
- Cases with PAD: Individuals with PAD

SUMMARY:
The goal of this study is to better understand how blood flows and how oxygen is utilized in the lower limbs of people who suffer from peripheral artery disease. This study will also assess how these factors affect treatment outcomes.

Specific aims include:

Aim 1: Utilize BB-NIR-DCS to differentiate PAD patients experiencing primary oxygen delivery limitations from those suffering from mitochondrial dysfunction.

Aim 2: Test the efficacy of BB-NIR-DCS at predicting individual responses to vascular intervention.

DETAILED DESCRIPTION:
Subjects that do not have peripheral artery disease will complete the study procedures up to two times (baseline and follow-up at 1-2 months).

Subjects diagnosed with peripheral artery disease may be asked to complete the study procedures up to 4 separate times (baseline, follow-up at 1-2 weeks, 1-2 months, and 4-6 months). The investigators will work with them to schedule each visit.

All participants will provide informed consent prior to participating in the study. The screening procedures will include collecting information about health history, age, sex, race/ethnicity, height, weight, and reasons one should not undergo an MRI or exercise.

The laboratory procedures will include questionnaires about quality of life and walking ability, Ankle- Brachial Index, functional performance measures (treadmill walking and six minute walk distance), wearable activity monitor and activity log, and lower limb MRI with muscle perfusion and oxygenation measures at rest and in response to physiologic provocation (ischemia-reperfusion and exercise).

Investigators may ask subjects to return on a separate day to repeat part, or all, of the study procedures depending on image quality and/or equipment performance.

ELIGIBILITY:
Inclusion Criteria:

* Cases, Aim 1

  1. 18 or older
  2. willing to participate under the conditions described in the informed consent form (ICF)
  3. eligible to sign the ICF
  4. established diagnosis of PAD confirmed by a physician
  5. able to comply with the study requirements
* Cases, Aim 2

  1) completed Aim 1
* Controls 1) asymptomatic, with no history or diagnosis of peripheral artery disease

Exclusion Criteria:

* Cases, Aim 1

  1. Ankle-Brachial Index >0.9 or <0.4
  2. isolated disease in aorta/iliac vessels
  3. unstable angina or myocardial infarction in past 12 months
  4. orthopedic or other physical limitations which would prevent data collection
  5. contraindications to MRI, including presence of a Pacemaker, presence of bone growth/ bone fusion stimulators, presence of tissue expander, presence of cochlear implants, unable to ambulate for 10 feet, receiving continuous Oxygen therapy, pregnancy, permanent Jewelry (screened using MRI safety screening form and verbal screening by MRI operator
* Cases, Aim 2

  1. unstable angina or myocardial infarction in past 12 months
  2. orthopedic or other physical limitations which would prevent data collection
  3. contraindications to MRI, including presence of a pacemaker, presence of bone growth/ bone fusion stimulators, presence of tissue expander, presence of cochlear implants, unable to ambulate for 10 feet, receiving continuous Oxygen therapy, pregnancy, permanent Jewelry (screened using MRI safety screening form and verbal screening by MRI operator).
* Controls 1) history of peripheral artery disease 2) overt cardiovascular disease (e.g. heart failure) 3) known pulmonary disease (excluding mild asthma) 4) current tobacco use 5) orthopedic or other physical limitations which would prevent data collection, 6) BP >150/90 mmHg at screening 7) contraindications to MRI, including presence of a pacemaker, presence of bone growth/ bone fusion stimulators, presence of tissue expander, presence of cochlear implants, unable to ambulate for 10 feet, receiving continuous Oxygen therapy, pregnancy, permanent Jewelry (screened using MRI safety screening form and verbal screening by MRI operator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases- 80 individuals with PAD.
  Controls- 40 healthy volunteers, of similar age, sex, and ethnicity as the PAD cases.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Quality of life | Baseline and up to 26 weeks
  Participants will complete a health questionnaire to gain a deeper understanding of their quality of life.
Ankle- Brachial Index | Baseline and upto 26 weeks
  The Ankle Brachial Index will be noninvasively assessed using the Smartdop XT device (Koven Technology, Inc.)
Walking ability | Baseline and upto 26 weeks
  Participants will complete a questionnaire to gain a deeper understanding of their walking ability
Functional performance | Baseline and upto 26 weeks
  Participants will be asked to walk as much as they can for six minutes (up and down a long hallway). Then, they will be asked to walk on a treadmill at 2 mph (3.2 km/h) at a grade of 10% for all as long as they can, or for a maximum of 10 minutes.
Steps taken | Baseline and upto 26 weeks
  Participants will be asked to wear an activity monitor on their wrist to track the number of steps they take each day for up to 6 months. A member of the study team will contact them by phone, email or text message each week to remind them to complete a log book of their daily activity.
Oxygen level of leg muscles | Baseline and upto 26 weeks
  Participants will be asked to perform exercise with their lower leg (affected leg, if they have peripheral artery disease) while they are in an MRI. A small plastic device (about the size of a match box) will also be placed on their lower limb. This device will measure the oxygen level of their leg muscles using near-infrared light.
Body composition | Baseline and up to 26 weeks
  An MRI will be performed across the upper and lower body to measure muscle size, muscle quality, adiposity and body structure.
Leg Exercise MRI | Baseline and upto 26 weeks
  Participants will be asked to perform exercise with their lower leg (affected leg, if they have peripheral artery disease) while they are in an MRI. The MRI will be used to measure the blood flow in leg and the oxygen level of the blood in their veins.
Lower Leg Ischemia-Reperfusion | Baseline and up to 26 weeks
  A blood pressure cuff will be inflated around the upper leg for 5 minutes before being released. Leg blood flow and vein oxygen saturation will be measured throughout.
Leg muscle size and quality | Baseline and up to 26 weeks
  An MRI of the leg will be performed to measure muscle size and tissue characteristics.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Texas at Arlington, Arlington, Texas
  - University of Texas Arlington, Arlington, Texas

IPD SHARING:
Plan to Share IPD: Undecided